CLINICAL TRIAL: NCT00851942
Title: Determination of Method-specific Normal Cortisol and Adrenal Hormone Responses to the Short Synacthen Test
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cardiff University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SPON 431-07
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Healthy; Adrenal Insufficiency; Hypopituitarism
Keywords: Volunteer; Hypoadrenalism; Hypopituitarism; Healthy volunteers
MeSH Terms: conditions — Adrenal Insufficiency; Hypopituitarism | interventions — Cosyntropin; adrenocorticotropin zinc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Synacthen 250 micrograms (Experimental): IV injection of 250 micrograms of Synacthen in 1m
  Interventions: Drug: Synacthen (Tetracosactrin)

INTERVENTIONS:
Drug: Synacthen (Tetracosactrin) — IV injection of 250 micrograms of Synacthen in 1ml
  Other Names: Synacthen

SUMMARY:
Objectives:

To establish valid serum total cortisol and salivary cut-offs for use with the short Synacthen test in patients with normal CBG concentrations.

To investigate, using current assays, the effect of assay differences on the serum total cortisol cut-off.

To explore the performance of these cut-offs in groups of patients with suspected adrenal insufficiency and high and low serum CBG concentration.

Methodology: An ACTH test (250 micrograms iv ACTH1-24) will be undertaken in healthy volunteers, women taking an oestrogen-containing oral contraceptive pill (OCP), patients with adrenal insufficiency and patients with low serum albumin. Serum cortisol in the samples collected from healthy volunteers will be measured using GC-MS, Advia Centaur (Siemens), Architect (Abbott), Modular Analytics E170 (Roche), Immulite 2000 (Siemens) and Access (Beckman) automated immunoassays. The estimated lower reference limit for the 30 min cortisol response to ACTH, defined as the 2.5th percentile of log-transformed concentrations, will be determined in this healthy population and used as a cut-off in the patient groups studied.

DETAILED DESCRIPTION:
Synacthen® is a synthetic analogue of ACTH which has been used since the 1960s to assess adrenal sufficiency. It is now well established as a first line test to investigate diseases of the hypothalamo-pituitary-adrenal axis and to assess adrenal function in patients on long-term corticosteroid therapy. Briefly, cortisol is measured before and after injection of 250 micrograms of Synacthen®. In a normal individual serum cortisol will rise to concentrations greater than an arbitrary value (typically 550 nmol/l) 30 minutes after administration of Synacthen®.

In 2004 the All Wales Clinical Biochemistry Audit group surveyed protocols for performing and interpreting short Synacthen® tests. This identified wide differences in practice within Wales. As a result standards were drawn up for performance of the test. It was noted that there was considerable variability or bias between cortisol immunoassays and that the cortisol cut-off chosen for interpretation of the short Synacthen® test should be method dependent.

Clark et al., in 1998 reported cortisol cut-offs following Synacthen® using 4 well established commercially available cortisol immunoassays. This study demonstrated considerable differences between the cortisol immunoassays used in clinical laboratories at the time. It was also apparent that there were differences in gender-related responses to Synacthen® although there was no dependence on age. In the 8 years since publication of this study there have been advances in formulation of cortisol immunoassays as well as the instrumentation used to perform analyses. At the University Hospital of Wales cortisol is currently assayed using the Bayer Centaur automated immunoassay analyser. This assay was not available at the time of the study by Clark et al.,. The investigators' current short Synacthen® test cut-offs therefore rely on historical reference ranges which have become outdated. A re-evaluation of the cortisol cut-off is required to ensure that patients are not incorrectly classified.

It has been long been recognised that oestrogens (including ethinyloestradiol prescribed in combined oral contraceptive pills) increase total (but not free) serum cortisol levels. The degree of increase is related to the dose used and is thought to be due to an elevation in cortisol binding globulin (CBG). However, no comparisons of total serum cortisol in response to Synacthen® have been performed between women taking oestrogens and those who are not. Knowledge of the salivary cortisol response may also be useful in patients with decreased serum CBG concentrations e.g. severe nephrotic syndrome in whom the serum cortisol response may be misleading. The investigators therefore plan to measure salivary cortisol as part of the investigators' study protocol to assess the response of free cortisol.

17 Hydroxyprogesterone (17OHP) is an intermediate in the biosynthesis of cortisol. Deficiency of 21-hydroxylase enzyme activity leads to an increased concentration of 17OHP in the peripheral circulation. The short Synacthen® test can be used to assist in diagnosis of mild cases of congenital adrenal hyperplasia. Current reference ranges are taken from the literature.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers will be in self-proclaimed good health
* Volunteers will be free of illness on the day of testing
* Volunteers will not be taking drug therapy.
* Patients will be free of intercurrent illness on the day of testing
* Patients will have a confirmed diagnosis of hypoadrenalism or hypopituitarism

Exclusion Criteria:

* Is pregnant or lactating. Females of childbearing potential must have a negative pregnancy test before enrollment onto the study. Non-child bearing potential is defined as post-menopausal for at least 1 year, surgical sterilisation or hysterectomy at least three months before the start of the study,
* Is using corticosteroids,
* has any significant intercurrent disease,
* has a history of thyroid or other autoimmune disease,
* has a previous history of hypersensitivity to Synacthen®,
* has a previous history of asthma
* has a history of allergic disorder
* has any mental condition rendering the patient unable to understand the nature or possible consequences of the study, and/or evidence of an uncooperative attitude.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2008-09; Primary Completion 2012-07-28 (Actual); Study Completion 2013-01-31 (Actual)

PRIMARY OUTCOMES:
The primary end-point of the study will be to establish method dependent cortisol cut offs for the normal response to Synacthen® using the 5th percentile. | Cortisol response at 30 minutes

SECONDARY OUTCOMES:
Cortisol measurements by immunoassay will be compared with the GC-MS gold standard method for normal volunteers and patients with hypopituitarism and hypoadrenalism. | Cortisol response at 30 minutes
Synacthen® responses in women taking ethinyloestradiol-containing contraceptive pills will be compared with those who are not. | Cortisol response at 30 minutes
We will establish cut offs for the salivary cortisol response to Synacthen® in normal volunteers using the 5th percentile. | Cortisol response at 30 minutes
We will establish a 17OHP cut off in response to Synacthen® in normal female volunteers using the 5th percentile. | 17OHP response at 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Aled Rees, MB BCh, PhD, Principal Investigator — Cardiff University
Locations (1):
- Clinical Research Facility, University Hospital of Wales, Cardiff, South Glamorgan, United Kingdom

REFERENCES:
- [Derived] Owen LJ, Adaway JE, Davies S, Neale S, El-Farhan N, Ducroq D, Evans C, Rees DA, MacKenzie F, Keevil BG. Development of a rapid assay for the analysis of serum cortisol and its implementation into a routine service laboratory. Ann Clin Biochem. 2013 Jul;50(Pt 4):345-52. doi: 10.1177/0004563212473448. Epub 2013 Jun 12. PMID 23761380